CLINICAL TRIAL: NCT04992949
Title: A Phase II Study of CPX-351 Monotherapy in Acute Myeloid Leukemia
Brief Title: Evaluation of CPX-351 Monotherapy in Acute Myeloid Leukemia Secondary to Myeloproliferative Neoplasm
Acronym: CPX-351 TA-SMP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Acute Leukemia French Association (Other); French Intergroup of Myeloproliferative syndromes (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPX-351 TA-SMP
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia; Myeloproliferative Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351

STUDY DESIGN:
Intervention Model Description: Open label multicenter phase II non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPX351 (Experimental): Induction : patients will receive induction treatment with CPX-351 100 U/m2 on days 1, 3, and 5. Patients who fail to achieve CR/CRi after the induction cycle will be offered a second induction course of CPX-351 100 U/m2 on days 1 and 3, at the investigators' discretion. If CR/CRi is not achieved following the second induction cycle, patients will go off study Consolidation : patients in CR/CRi after induction cycle will receive up to 2 course of CONSOLIDATION therapy with CPX-351 65 U/m2 on days 1 and 3. CPX351 doses could be reduced to 65 U/m2 on day 1 in case of unacceptable toxicity following the previous course.
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — Induction : patients will receive induction treatment with CPX-351 100 U/m2 on days 1, 3, and 5. Patients who fail to achieve CR/CRi after the induction cycle will be offered a second induction course of CPX-351 100 U/m2 on days 1 and 3, at the investigators' discretion. If CR/CRi is not achieved following the second induction cycle, patients will go off study
  Consolidation : patients in CR/CRi after induction cycle will receive up to 2 course of consolidation therapy with CPX-351 65 U/m2 on days 1 and 3. CPX351 doses could be reduced to 65 U/m2 on day 1 in case of unacceptable toxicity following the previous course.
  Allo-SCT : patients for whom an allo-SCT is planned will receive a maximum of one consolidation cycle

SUMMARY:
The three classic myeloproliferative neoplasms (MPNs) include polycythemia Vera (PV), essential thrombocythemia (ET) and primary myelofibrosis (PMF). The natural history of these MPNs is the possible progression to acute myeloid leukemia (MPN-blast phase) at variable percentage depending the entity. Leukemic transformation of MPN occurs in 8% to 23% of primary myelofibrosis (PMF) patients in the first 10 years after diagnosis and in 4% to 8% of polycythemia vera (PV) and essential thrombocytosis (ET) patients within 18 years after diagnosis. The risk for leukemic transformation is increased by exposure to cytotoxic chemotherapy. The molecular pathogenesis of MPN-blast phase remains an area of active research.

The prognosis of blast phase MPNs is very poor : approximately 50% of the patients are deemed eligible for intensive treatment (ie. conventional induction chemotherapy regimen with anthracyclines and cytarabine). The patients who are not fit for such intensive treatment approach due to age or comorbidities, are treated with Hypomethylating agents, low dose palliative chemotherapy, or supportive care. Nevertheless, there is a need for more effective and better tolerated treatment approaches in order to increase the response rate and hence, the transplant rates which should translate into improved survival.

CPX-351 is a new formulation of cytarabine and daunorubicin encapsulated at a fixed 5:1 molar-ratio in liposomes that exploits molar ratio-dependent drug-drug synergy to enhance antileukemic efficacy.

Based on similarities between post-myelodysplastic syndrome (MDS) and post-MPN secondary AML in terms of disease resistance to chemotherapy, of fragile patient profile, The hypotheses made is that CPX-351 may improve the results of induction chemotherapy without increasing its toxicity and therefore may increase the proportion of patients who could benefit from an allogeneic Stem Cell Transplantation (SCT).

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the Complete Remission (CR/CRi) rate after treatment with CPX-351 in patients with AML secondary to myeloproliferative neoplasms (post-MPN AML).

The hypotheses made is that treatment with CPX-351 will improve the historical response rate from 45% to 65%. The exact single stage Phase II design was used to calculate the number of patients. The null hypothesis H0 is that the probability p of CR/CRi rate with CPX351 is equal or lower than the historical rate p0 of 45% (H0: p≤p0). The alternative hypothesis H1 that is p>p0, supposing that CR/CRi rate will be 65% using CPX351. Considering an alpha risk of 5% and a power of 80%, 42 patients will be included, and H0 will be rejected if at least 25 patients achieve CR /CRi (R-project, "clinfun" package).

Inclusion period : 36 months

Treatment period (6 months) :

* one or two cycles of induction treatment with CPX-351 (depending on CR/CRi achieving). If CR/CRi is not achieved following the induction phase, patients will go off study.
* 2 courses of consolidation therapy with CPX-351 (patients for whom an allo-SCT is planned will receive a maximum of one consolidation cycle)

All included patients will be followed for 60 days after the End of Treatment (EOT) or at the date of allogeneic stem cell transplantation when appropriate : the day-60 follow-up visit will be the End Of Study (EOS) visit. The anti-leukemic chemotherapy administrated after relapse will be recorded.

After completion of the study, subjects will be followed-up at regular intervals (every 3 months) to collect information on the subjects' survival and disease (relapse) status. Survival status will be collected until death, or withdrawal of consent or lost to follow-up, whichever occurs first..

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of newly secondary AML according to WHO 2016 classification following an antecedent of Myeloproliferative Neoplasm including Essential Thrombocythemia (ET), Polycythemia Vera (PV), primary or secondary Myelofibrosis
* Performance status 2 Eastern Cooperative Oncology Group (ECOG) grading.
* Eligible for standard intensive chemotherapy
* Absence of concomitant severe cardiovascular disease which would make intensive chemotherapy impossible, i.e. arrhythmias requiring chronic treatment, congestive heart failure or symptomatic ischemic heart disease, reduced left ventricular function assessed by multigated acquisition (MUGA) scan or echocardiogram. Cardiac ejection fraction ≥ 50% by echocardiography ou MUGA
* Patient must have adequate organ function as indicated by the following laboratory values:

  * Renal

    * Serum creatinine: < 2 mg/dl OR calculated creatinine clearance*: ≥ 30 mL/min by MDRD formula for patients with creatinine levels > 1.5 X institutional Upper Limit Normal (ULN)
  * Hepatic

    * Serum total bilirubin: ≤ 2.5 X ULN OR direct bilirubin ≤ ULN for patients with total bilirubin levels ≥ 2 mg/dL unless Gilbert's Syndrome
    * Aspartate-Amino-Transferase (ASAT) and Alanine-Transaminase (ALAT): ≤ 2.5 times ULN
    * Alkaline Phosphatase: ≤ 5 X ULN, if > 2.5 X ULN, then liver fraction should be ≤ 2.5 X ULN *Creatinine clearance should be calculated per institutional standard
* Life expectancy should be of 12 weeks at least according to investigator evaluation
* Female patients of childbearing potential must have a negative serum pregnancy test (β-hCG) within 72 hours prior to receiving the first dose of CPX-351. Female patients who are not post-menopausal, free from menses for > 2 years or surgically sterilized, will have to use adequate barrier methods of contraception to prevent pregnancy or agree to abstain from becoming pregnant throughout the study, starting with Visit 1.
* Male patients agree to use an adequate method of contraception for the duration of the study. Men should be advised not to father a child while receiving CPX-351 and for 3 months post study.
* Patients have the ability to understand and willingness to sign an informed consent form indicating the investigational nature of the study.

Exclusion Criteria:

* MPN/MDS mixed types
* Prior therapy for AML transformation except for Hydroxyurea
* Prior treatment with growth factors such as erythropoietin alfa (EPO) or granulocyte colony-stimulating factor (G-CSF), low-dose oral chemotherapy or Hypomethylating agents chemotherapy given in the chronic phase of MPN in the 30 days before inclusion, except for hydroxyurea.
* Uncontrolled undercurrent illness or circumstances that could limit compliance with the study, including but not limited to the following: symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, pancreatitis, or psychiatric or social conditions that may interfere with patient compliance.
* Active and uncontrolled infection
* Current participation or participation in a study with an investigational compound or device within 30 days of initial dosing with study drug
* Patients with acute promyelocytic leukemia.
* Known human immunodeficiency virus (HIV) infection or HIV-related malignancy
* Clinically active hepatitis B or hepatitis C infection.
* Known allergy or hypersensitivity to any component of CPX-351.
* Currently active second malignancy, other than non-melanoma skin cancer and in situ carcinoma of the cervix. Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >3 years or are considered by their physician to be at less than 30% risk of relapse
* Clinical evidence of Central Nervous System Leukemia.
* Pregnancy or breastfeeding during the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Rate of CR/CRi after first induction therapy | After 28 to 42 days after one cycle of 5 days of CPX351
  Rate of CR/CRi according to ELN2017 criteria
Rate of CR/CRi after second induction therapy | If applicable, after 28 to 31 days after a second cycle of 3 days of CPX351
  Rate of CR/CRi according to ELN2017 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme REY, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (34):
- France (34):
  - AMIENS - CHU Amiens Picardie, Amiens
  - ANGERS - CHU - Maladies du sang, Angers
  - AVIGNON - Centre Hospitalier, Avignon
  - BAYONNE - CH de la Côte Basque - Hématologie, Bayonne
  - AVICENNE - Centre de Recherche Clinique, Bobigny
  - BREST - Hôpital Morvan, Brest
  - CAEN - CHU Caen - IHBN, Caen
  - CLAMART - Hôpital d'Instruction des Armées de Percy, Clamart
  - Clermont-Ferrand - Chu Estaing, Clermont-Ferrand
  - CRETEIL - CHU Henri Mondor, Créteil
  - Grenoble - CHUGA - Hématologie Clinique, Grenoble
  - LILLE CHU - Hôpital Claude Huriez, Lille
  - LIMOGES - CHU Dupuytren 1, Limoges
  - LYON-Centre Léon Bérard, Lyon
  - MARSEILLE - Institut Paoli-Calmettes, Marseille
  - MONTPELLIER - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - NANTES - Hôpital Hôtel Dieu - Hématologie Clinique, Nantes
  - NICE - Centre Antoine Lacassagne, Nice
  - NICE - CHU - Hopital Archet 1, Nice
  - NIMES - CHU Caremeau, Nîmes
  - ORLEANS - CHR - Hématologie, Orléans
  - Paris St Antoine, Paris
  - Paris Saint Louis, Paris
  - BORDEAUX - Hôpital Haut-Levêque, Pessac
  - LYON HCL - CH Lyon Sud, Pierre-Bénite
  - POITIERS - Hôpital La Milétrie - Hématologie Clinique, Poitiers
  - REIMS - Hôpital Robert Debré - Hématologie Clinique, Reims
  - RENNES - Hôpital Pontchaillou - Hématologie, Rennes
  - Strasbourg - Icans, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - TOURS - Hôpital Bretonneau, Tours
  - NANCY - CHU de Brabois, Vandœuvre-lès-Nancy
  - VERSAILLES - Hôpital André Mignot, Versailles
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Courtier F, Carbuccia N, Garnier S, Guille A, Adelaide J, Cervera N, Gelsi-Boyer V, Mozziconacci MJ, Rey J, Vey N, Chaffanet M, Birnbaum D, Murati A. Genomic analysis of myeloproliferative neoplasms in chronic and acute phases. Haematologica. 2017 Jan;102(1):e11-e14. doi: 10.3324/haematol.2016.152363. Epub 2016 Oct 14. No abstract available. PMID 27742771
- [Background] Luque Paz D, Jouanneau-Courville R, Riou J, et al. Leukemic evolution of polycythemia vera and essential thrombocythemia: genomic profiles predict time to transformation. Blood Adv. 2020;4(19):4887-4897. Blood Adv. 2020 Nov 24;4(22):5651. doi: 10.1182/bloodadvances.2020003711. No abstract available. PMID 33206963